CLINICAL TRIAL: NCT00216944
Title: Balanced Anesthesia for Intubation of Newborn Premature Infants - a Randomized Intervention Study
Brief Title: Balanced Anesthesia for Intubation of Premature Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Vineta Fellman/Proffessor, Department of Peadiatrics, Lund University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUDRACT EU 2004-001583-52
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-12

CONDITIONS: Premature Birth
Keywords: Intubation; premedication
MeSH Terms: conditions — Premature Birth | interventions — Intubation, Intratracheal; Respiratory Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Premedication with atropine and morphine
  Interventions: Procedure: Tracheal intubation for respiratory care in preterm infants
- 2 (Active Comparator): Premedication with glycopyrronium, thiopental, suxamethonium and remifentanil
  Interventions: Procedure: Tracheal intubation for respiratory care in preterm infants

INTERVENTIONS:
Procedure: Tracheal intubation for respiratory care in preterm infants — Premedication with atropine 0.02 mg/kg and morphine 0.03 mg/kg
  Arms: 1
Procedure: Tracheal intubation for respiratory care in preterm infants — Premedication with glycopyrronium 0.005 mg/kg, thiopental 2-3 mg/kg (< 2 kg 2 mg/kg), suxamethonium 2 mg/kg and remifentanil 0.001 mg/kg
  Arms: 2

SUMMARY:
The study aim is to compare a balanced anesthesia of the medicines used in all other age groups with the routine premedication in use for premature's with regards to the success in the intubation procedure, the need for analgesia during and after intubation and the stress reaction. In addition a pain scale for prolonged stress/pain for premature neonates in NICU-care will be validated, and the individual pharmacogenetic profile in relation to the need of morphine after the intubation will be investigated. The hypothesis is that balanced anesthesia before intubation facilitates the procedure, decreases the amount of stress and pain related to it, and causes a decreased need for analgesia after the intubation.

ELIGIBILITY:
Inclusion Criteria:

* <37 gw at birth
* <72 hours postnatal age, not previously intubated and no analgetics or sedatives the last 12 hours or >72 hours postnatal age, primary or reintubation
* Informed consent from parents

Exclusion Criteria:

* Intubation directly postnatally at the delivery room
* Asphyxia (apgar <4 at 10 min, Umb-pH <7,0
* S-Potassium > 6,5
* Major malformations
* Postsurgery intubation
* Included in an other intervention study first week in life
* Other intervention study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Success of intubation according to a specific score including duration of the procedure and changes in oxygen saturation, blood pressure and heart rate during the intubation | 6-9 months

SECONDARY OUTCOMES:
Pain score at intubation | 6-9 months
Biochemical stress/pain response | 6-9 months
Physiological stress/pain response | 6-9 months
Behavioural stress/pain response | 6-9 months
Neurophysiological stress/pain response (aEEG) | 6-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Vineta Fellman, Professor, Principal Investigator — Lund University and Lund University Hospital
Locations (1):
- Neonatal Departement Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Norman E, Wikstrom S, Rosen I, Fellman V, Hellstrom-Westas L. Premedication for intubation with morphine causes prolonged depression of electrocortical background activity in preterm infants. Pediatr Res. 2013 Jan;73(1):87-94. doi: 10.1038/pr.2012.153. Epub 2012 Nov 5. PMID 23128421
- [Derived] Norman E, Wikstrom S, Hellstrom-Westas L, Turpeinen U, Hamalainen E, Fellman V. Rapid sequence induction is superior to morphine for intubation of preterm infants: a randomized controlled trial. J Pediatr. 2011 Dec;159(6):893-9.e1. doi: 10.1016/j.jpeds.2011.06.003. Epub 2011 Jul 27. PMID 21798556